CLINICAL TRIAL: NCT01234597
Title: A Comparative Study to Evaluate the Prandial Treatment Adjustment Effect Via Continuous Glucose Monitoring on Type 2 DM Patients Uncontrolled With a Basal Insulin or Premix Once a Day
Brief Title: Evaluation of the Prandial Treatment Adjustment Effect Via Continuous Glucose Monitoring on Type 2 Diabetes Mellitus (DM) Patients Uncontrolled With a Basal Insulin or Premix Once a Day
Acronym: SeLan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_05146; U1111-1116-2926 (Other: UTN)
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; insulin glulisine

ARMS (2):
- Arm A: Without Continous Glucose Monitoring (CGM) sensor (Active Comparator): Run-in phase: insulin glargine is administered at initial dosage according to FBG measurements performed by the patient by using a glucometer .
  Treatment phase: insulin glulisine is administered at initial dosage according to FBG measurements performed by the patient by using a glucometer. Then, adjustment of the dosage is performed by the treating physician
  Interventions: Drug: INSULIN GLARGINE (HOE901); Drug: INSULIN GLULISINE (HMR1964)
- Arm B: Continous Glucose Monitoring (CGM) sensor (Experimental): Run-in phase: insulin glargine is administered at initial dosage according to FBG measurements performed by the patient by using a glucometer .
  Treatment phase: the patients are connected to a CGM sensor. Insulin glulisine is administered at initial dosage according to FBG measurements performed by the patient by using a glucometer. Then, adjustment of the dosage is performed by the national coordinator based on the data collected in the past previous days of CGM sensor monitoring.
  Interventions: Drug: INSULIN GLARGINE (HOE901); Drug: INSULIN GLULISINE (HMR1964)

INTERVENTIONS:
Drug: INSULIN GLARGINE (HOE901) — Pharmaceutical form: solution for injection Route of administration: subcutaneous
Drug: INSULIN GLULISINE (HMR1964) — Pharmaceutical form:Solution for injection Route of administration: Subcutaneous

SUMMARY:
Primary Objective:

To evaluate the effect of prandial treatment adjustment, based on continuous blood glucose monitoring, on glucose control in type 2 diabetes patients who are not controlled by treatment with once daily basal insulin or mixed insulin, requiring treatment with basal plus regimen

DETAILED DESCRIPTION:
The study duration for each patient is 24 weeks +/- 1 week broken down as follows:

* Run-in phase: 8 weeks
* Follow - up Period: 16 weeks

The maximal possible time window during the study is +/- one week throughout the study.

ELIGIBILITY:
Inclusion criteria:

Run-in period:

1. Type 2 diabetes
2. HbA1c≥ 8.5% (in a test of the last month)
3. Age above 21 years
4. Patients continuously treated with basal insulin or mixed insulin once daily for the last 6 months
5. Signed informed consent form
6. Patients who according to their physician are eligible to the study

Randomization:

1. HbA1c > 7.5%
2. FPG < 130 mg/dl

Exclusion criteria:

1. Type 1 diabetes
2. Patients continuously treated with short-acting insulin or mixed insulin more than once daily for 3 weeks during the last 6 months.
3. Pregnant or breastfeeding women.
4. Patients with allergy to insulin.
5. Patients with severe diseases characterized by recurrent hospitalizations, including: Severe renal insufficiency, severe cardiac insufficiency, active oncological disease or oncological disease requiring chemotherapy.
6. Patients with mobility difficulties and/or difficulties communicating with the investigator

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2012-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Changes in Hemoglobin A1c (HbA1c) level | Baseline, week 24

SECONDARY OUTCOMES:
Rate of hypoglycemia | Week 24
Changes in insulin glargine dose | Baseline, week 24
Changes in insulin glulisine dose | Baseline, week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (11):
- Israel (11):
  - Investigational Site Number 376003, Beersheba
  - Investigational Site Number 376007, Haifa
  - Investigational Site Number 376004, Kfar Saba
  - Investigational Site Number 376012, Lod
  - Investigational Site Number 376013, Nazareth
  - Investigational Site Number 376006, Netanya
  - Investigational Site Number 376001, Ramat Gan
  - Investigational Site Number 376009, Sakhnin
  - Investigational Site Number 376008, Tel Aviv
  - Investigational Site Number 376010, Tel Aviv
  - Investigational Site Number 376011, Tel Aviv